CLINICAL TRIAL: NCT01859897
Title: A Prospective Multicenter Study to Evaluate Usefulness of Cardio-Ankle Vascular Index in Japan
Acronym: CAVI-J
Status: Completed | Type: Observational
Sponsor: CAVI-J Study Group (Other)
Collaborators: Toho University (Other); Ehime University Graduate School of Medicine (Other); Dokkyo Medical University (Other); Okayama University (Other)
Responsible Party: Sponsor-Investigator, CAVI-J Study Group, CAVI-J study Group, Okayama University
Organization: Okayama University (Other)
Other Study IDs: okayama-1692
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Stroke; Cardiovascular Death; Nonfatal Myocardial Infarction
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Optimal therapy: All subjects will be treated by optimal medical therapy and lifestyle modification.

SUMMARY:
The objective of this five-year prospective observational follow-up study is to examine the additional benefits of using cardio-ankle vascular index (CAVI) as a predictive indicator of cardiovascular events in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

Patients between 40 and 74 years of age who have either of the following:

1. Type 2 diabetes mellitus
2. Metabolic syndrome
3. Grade I to III hypertension with the third layer of risk factors according to the guidelines for the management of hypertension japanese society of hypertension(JSH)2009
4. Chronic kidney disease(stage G3a or G3b) according ot the clinical Practice Guidebook for Diagnosis and Treatment of Chronic Kidney Disease 2012 in Japan
5. History of coronary artery disease or noncardiogenic cerebral infarction

Exclusion Criteria:

1. Under 40 years of age or over 74 years of age
2. An ankle-brachial index less than 0.9
3. Chronic atrial fibrillation
4. Current symptoms of heart failure(NYHA class III or IV) or left ventricular dysfunction (EF below 40%)
5. Malignancy
6. Chronic kidney disease(G4 or G5)according ot the clinical Practice Guidebook for Diagnosis and Treatment of Chronic Kidney Disease 2012 in Japan
7. chronic dialysis due to renal failure
8. Taking steroids/immunosuppressants
9. Hepatocirrhosis

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primiary care clinic and hospital
Sampling Method: Non-Probability Sample
Enrollment: 3026 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
major cardiac events | five years
  cardiac death, nonfatal myocardial infarction, stroke

SECONDARY OUTCOMES:
all cause mortality, cardiovascular events, and renaly dysfunction | five years
  all cause death, angina pectoris (with revascularization), New incidence of lower limb peripheral arterial disease(including lower limb arteriosclerosis obliterans), Aortic aneurysm, Aortic dissection, Heart failure that requires hospitalization, Deterioration in renal function (dialysis or renal transplantation)

OTHER OUTCOMES:
Change in CAVI and cardiovascular events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hajime Orimo, MD, Principal Investigator — Kenkoin Clinic
Locations (1):
- Okayama University, Okayama, Japan

REFERENCES:
- [Derived] Miyoshi T, Ito H, Shirai K, Horinaka S, Higaki J, Yamamura S, Saiki A, Takahashi M, Masaki M, Okura T, Kotani K, Kubozono T, Yoshioka R, Kihara H, Hasegawa K, Satoh-Asahara N, Orimo H; CAVI-J (Prospective Multicenter Study to Evaluate Usefulness of Cardio-Ankle Vascular Index in Japan) investigators *. Predictive Value of the Cardio-Ankle Vascular Index for Cardiovascular Events in Patients at Cardiovascular Risk. J Am Heart Assoc. 2021 Aug 17;10(16):e020103. doi: 10.1161/JAHA.120.020103. Epub 2021 Aug 7. PMID 34369198